CLINICAL TRIAL: NCT02200198
Title: Effect of Respiratory Muscle Training in Malnourished Patients Undergoing Upper Abdominal Surgery
Brief Title: Respiratory Muscle Training in Malnourished Patients Undergoing Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0613/07
Record Dates: First submitted 2014-07-23; First posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Undernutrition; Surgery
Keywords: undernutrition; abdominal surgery; respiratory muscles; muscles strength; pulmonary complication; perioperative care
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Inspiratory group (Active Comparator): Inspiratory muscle training
  Interventions: Other: Inspiratory muscle training
- Sham group (Sham Comparator): Sham training
  Interventions: Other: Sham group
- Expiratory group (Experimental): Expiratory muscle training
  Interventions: Other: Expiratory muscle training

INTERVENTIONS:
Other: Expiratory muscle training — Patient performs training for 30 minutes per day, during 7 consecutive days, using a Threshold with Positive Expiratory Pressure with a load of 30% of maximal expiratory pressure assessed by digital peak respiratory pressure monitor
  Arms: Expiratory group
Other: Inspiratory muscle training — Patient performs training for 30 minutes per day, during 7 consecutive days, using a Threshold for Inspiratory Muscle Training with a load of 30% of maximal inspiratory pressure assessed by digital peak respiratory pressure monitor
  Arms: Inspiratory group
Other: Sham group — Patient performs training for 30 minutes per day, during 7 consecutive days, using a Threshold without load
  Arms: Sham group

SUMMARY:
Malnutrition affects 50% of hospitalized patients around the world and causes changes in respiratory muscles predisposing the development of pulmonary complications probable, because of the ineffectiveness of cough. How the training of respiratory muscles can improve the effectiveness of cough, malnourished patients could benefit from this train however, the training of the muscles in malnourished patients has not been tested for safety or efficiency. So, the aim of this study is to assess the safety and efficiency of respiratory muscle training to improve the potency of cough in malnourished patients.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized malnourished patients (BMI ≤ 20 Kg/m2, loss of body weight ≥ 10% unintentional, or serum albumin <3.5 g/dL)
* candidate to elective abdominal surgery
* ability to perform all evaluations and training

Exclusion Criteria:

* previous respiratory disease
* necessity of over than 48h of mechanical ventilation
* reoperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Expiratory peak flow in spirometry | on the 8th day of protocol (after 7 dyas of training)
  Assessed as expiratory peak flow in spirometry

SECONDARY OUTCOMES:
Maximum respiratory pressures | on the 8th day of protocol (after 7 days of training)
  Assessed by digital peak respiratory pressure monitor as maximum inspiratory pressure and maximum expiratory pressure
Postoperative pulmonary complication | participants will be followed for the duration of hospital stay after surgery, an expected average of 10 days
  The following pulmonary complications were considered: atelectasis with clinical consequences, hypoxemia with oxygen saturation <85%, and need for supplemental oxygen, pneumonia and acute respiratory failure.
  The diagnosis of complication was performed by a physician who was blinded to the intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Celso RF Carvalho, PhD, Study Director — University of Sao Paulo
Locations (1):
- Hospital of Clinics of Sao Paulo, São Paulo, São Paulo, Brazil